CLINICAL TRIAL: NCT04412317
Title: National Observatory of the Care of Young Sick Children in Community or Not, Indications and Cost-effectiveness of PCR-Sars-CoV-2 - VIGIL Study
Brief Title: Use of PCR-Sars-CoV-2 in Children
Acronym: VIGIL
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Intercommunal Creteil (Other)
Collaborators: Association Clinique Thérapeutique Infantile du val de Marne (Other); Groupe de Pathologies Infectieuses Pédiatriques (GPIP) (Other); AFPA (Unknown); Francophone Pediatric Resuscitation and Emergency Group (GFRUP) (Other)
Responsible Party: Sponsor
Other Study IDs: VIGIL
Record Dates: First submitted 2020-05-30; First posted 2020-06-02 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Covid-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children < 15 years old: Patients under 15 years old who consults a physician on an outpatient basis or in the emergency room and who requires a Sars-CoV-2 RT- PCR (nucleic acid using real-time reverse-transcriptase polymerase-chain-reaction) diagnostic

SUMMARY:
The VIGIL study was set up at the beginning of the pandemic, in the spring of 2020, at a time when diagnostic testing for SARS-CoV-2 had to be performed according to specific clinical criteria (even if no clinical picture suggestive of COVID had been clearly identified). The management of sick young children (with respiratory tract infection that could be attributed to COVID) by pediatricians (infectious diseases specialists, emergency physicians, general practitioners, and outpatients) was facilitated by an algorithm whose objective was to help define the indications for SARS-CoV-2 PCR and subsequently for antigenic testing. The current technique of deep nasopharyngeal swabbing (for PCR or antigenic testing) is delicate and difficult in children, and is therefore a serious handicap for community-based screening, especially since infectious episodes are frequent in children. Since then, nasal self-tests that can be easily used in children have been commercialized and have facilitated screening.

Because of the similarity between the clinical signs of respiratory tract infections in children, it is often impossible to distinguish between different viral respiratory infections and epidemics may overlap in time. However, the identification of the pathogen is the key to improve management of these infectious diseases. The VIGIL study is therefore continuing, still facilitated by the existence of an active pediatric network existing for 20 years. ACTIV AFPA and GPIP have created networks of hospital and ambulatory pediatricians who actively participate in various observatories https://www.jpeds.com/article/S0022-3476(17)31606-2/fulltext To date, these observatories have resulted in the publication of more than 80 articles in international journals (https://www.activ-france.com/fr/publications).

ELIGIBILITY:
Inclusion Criteria:

* Children under 15 years of age
* Prescription of a PCR-Sars-CoV-2
* VIGIL information note given to parents

Exclusion Criteria:

* Refusal to participate by the patient, family member or legal representative (depending on the situation)

Max Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Child from birth to 14 years of age consulting their doctor
Sampling Method: Non-Probability Sample
Enrollment: 12000 (Estimated)
Dates: Start 2020-06-03 (Actual); Primary Completion 2024-05-30 (Estimated); Study Completion 2024-05-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of children screened with a positive PCR result or a positive Rapid Antigenic Diagnostic (RAD) test | At inclusion
  Number of positive PCR result or a positive Rapid Antigenic Diagnostic (RAD) test on total number of PCR

SECONDARY OUTCOMES:
Number of symptomatic children | the day of PCR or RAD result
  Number of positive PCR result in the sick child in the presence of a Covid contagion in the family environment or not on total number of PCR
presence or absence of positive people in close contacts | the day of PCR or RAD result
  Number of RAD-Sars-CoV-2 positive in the sick child in the presence of a Covid contagion in the family environment or not on number of negative RAD-Sars-CoV-2
Percentage of RAD RSV and Flu positive in children with respiratory tract infection | the day of PCR or RAD result
  Number of RAD RSV and Flu positive in children with respiratory tract infection on total number of tests
Accuracy of antigen test compared to PCR | the day of PCR or RAD result
  Sensibility and specificity of the test

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - ACTIV network, Créteil
  - PARI network, Créteil

REFERENCES:
- See also: From the original SARS-CoV-2 strain to the Omicron variant: Predictors of COVID-19 in ambulatory symptomatic children — https://pubmed.ncbi.nlm.nih.gov/36116761/
- See also: Diagnostic accuracy of SARS-CoV-2 rapid antigen test from self-collected anterior nasal swabs in children compared to rapid antigen test and RT-PCR from nasopharyngeal swabs collected by healthcare workers: A multicentric prospective study — https://pubmed.ncbi.nlm.nih.gov/36210936/
- See also: Assessment of SARS-CoV-2 testing in children during a low prevalence period (VIGIL study 1) — https://pubmed.ncbi.nlm.nih.gov/34271254/